CLINICAL TRIAL: NCT02534857
Title: A Randomized Double Blinded Controlled Study Comparing a Shorter Exposure of Oocyte to Spermatozoa Versus a Standard Incubation on the Live Birth Rate of In-vitro Fertilization Treatment
Brief Title: A Study Comparing a Shorter Exposure of Oocyte to Spermatozoa Versus a Standard Incubation on the Live Birth Rate of In-vitro Fertilization Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, chen zhi qin, Shanghai First Maternity and Infant Hospital, Shanghai First Maternity and Infant Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ShanghaiFMIH
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Fertility; In Vitro Fertilization
Keywords: randomized double blinded study; live birth rate; IVF treatment; brief incubation of oocytes and sperm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental): Those allocated to the intervention arm, all the oocytes will be exposed to spermatozoa for 2 hours and gently wash through two organ dishes containing 1.5 ml of equilibrated medium, and then transferred to the corresponding microdroplet of equilibrated fresh medium. Surrounding cumulus cell will be retained, not removed from the ooctyes.
  Interventions: Procedure: a shorter exposure of oocyte to spermatozoa
- Control arm (Placebo Comparator): Women who allocated to the control arm, all the oocytes will be exposed to spermatozoa for 20 hours, and checked for fertilization on day 1 (20 hours) after denuding
  Interventions: Procedure: a shorter exposure of oocyte to spermatozoa

INTERVENTIONS:
Procedure: a shorter exposure of oocyte to spermatozoa — Shorter exposure of oocyte to spermatozoa group: oocytes will be exposed to spermatozoa for 2 hours
  Other Names: brief co-incubation insemination

SUMMARY:
In vitro fertilization (IVF) treatment is now commonly used to treat infertile couples. During IVF treatment, oocytes and sperm are routinely incubated overnight and this may lead to suboptimal culture conditions because of increased reactive oxygen species (ROS) produced by sperm in the standard incubation. High levels of ROS can adversely affect the quality of the embryos, result in hardening of the zona pellucida and impair the implantation capacity of embryos. Studies shows successful fertilization of an oocyte occurs 20mins after the gametes are put together. Sperm can penetrate through the cumulus cells within 15min, and 80% of oocytes can be fertilized when they are exposed to a large number of spermatozoa within 1hr. As an attempt to avoid possible detrimental effects on the oocytes from long exposure to sperm, the brief incubation insemination protocol was developed. It implies that prolonged incubation of oocytes and sperm may not be necessary and may even be harmful. Some reports suggest that a sperm-oocyte exposure time of 1-6 h improves IVF outcomes. However, other studies report no such advantage with a short insemination time .

A recent meta-analysis shows brief incubation of gametes was associated with significantly higher rates of clinical pregnancy , ongoing pregnancy and higher rate of implantation than standard incubation. But the rates of normal fertilization, good quality embryos and polyspermy were not significantly different compared with standard incubation. In a Cochrane meta-analysis, eight RCTs with 733 women were included, and showed similar results. But it only reported clinical pregnancy rate and ongoing pregnancy rate which were significantly higher in brief incubation group than standard incubation. However, the live birth rate, which is the important outcome parameter, was not reported in all these studies. It is uncertain whether brief incubation improves the life birth rate compared with standard incubation.

The aim of this randomized double blinded study is to compare the live birth rate of IVF treatment following brief incubation of oocytes and sperm versus standard incubation. The hypothesis is that a brief incubation improves the live birth rate of IVF treatment.

DETAILED DESCRIPTION:
1. Background

   In vitro fertilization (IVF) technique is now commonly used for the treatment of infertile couples. To obtain better outcomes of IVF, it is important to enhance embryo quality by optimizing IVF techniques. In IVF procedures, oocytes and sperm are routinely co-incubated overnight, which may expose oocytes and zygotes to suboptimal culture conditions with increased reactive oxygen species (ROS) produced by sperm in this long term culture[1]. High levels of reactive oxygen species (ROS) can adversely affect the quality of the embryos, result in hardening of the zona pellucida and impair the implantation capacity of embryos [2-4]. Studies shows successful fertilization of a mamamal oocyte occurs 20mins after gametes meet [5]. Sperm can penetrate through the cumulus cells within 15min, and 80% of oocytes can be fertilized when they are exposed to a large number of spermatozoa within 1hrs[1]. As an attempt to avoid possible detrimental effects on the oocytes from long exposure to sperm, the brief co-incubation insemination protocol was developed. It implies that long-term co-incubation of oocytes and sperm may not be necessary and may even be harmful. Some reports suggest that a sperm-oocyte exposure time of 1-6 h improves IVF outcomes[1,2,6,7] However, other studies report no such advantage with a short insemination time[8,9,10] .

   Recent published Meta analysis shows[11] brief co-incubation of gametes was associated with significantly higher rates of clinical pregnancy (RR: 1.84, 95% CI: 1.24-2.73), ongoing pregnancy (RR: 1.73, 95%CI: 1.27-2.33) and higher rate of implantation (RR: 1.80, 95% CI: 1.43-2.26) than standard insemination. But the rates of normal fertilization (RR: 0.98, 95% CI: 0.93-1.02), good quality embryos (RR: 1.24, 95% CI: 1.0-1.53) and polyspermy (RR: 0.84, 95% CI: 0.7-1.01) were not significantly different compared with standard insemination. In another Cochrane meta-analysis[12] eight RCTs with 733 women were included, and got the similar results. But it only reported clinical pregnancy rate, ongoing pregnancy rate which was significantly higher in brief co-incubation group than standard insemination. For the miscarriage rate, there were six miscarriages in one trial including 167 women. This low quality evidence suggested no significant difference in the odds of miscarriage between brief co-incubation and standard insemination (OR 1.98, 95% CI 0.35 to 11.09; P = 0.44). And live birth was not reported in the included studies, it is unclear whether brief co-incubation improves the life birth rate compared with the standard overnight insemination protocol.

   Drawbacks inherent to the quality of these studies, such as lack of allocation concealment and no blinding, limit the quality of the available evidence. To better evaluate these issues, more well designed RCTs are required to assess whether brief co-incubation would contribute to a higher live birth rate and a lower miscarriage rate compared to the standard overnight insemination protocol.
2. Objectives:

   The objective of the present randomized, double blinded controlled study is to compare clinical effectiveness (especially on live birth rate) of a shorter exposure of oocyte to spermatozoa compared to a standard incubation in women undergoing IVF treatment.
3. Trial design:

A total of 280 infertile women undergoing IVF treatment will be randomized into one of the following two groups by computer-generated random numbers that was placed in sealed envelopes:

Shorter exposure of oocyte to spermatozoa group: oocytes will be exposed to spermatozoa for 2 hours Standard incubation group: oocytes will be exposed to spermatozoa for 20 hours

Treatment of subjects

All techniques of IVF including ovarian stimulation will be according to local protocols.

4.1 Ovarian stimulation and IVF

All women started their IVF treatment with ovarian stimulation using either the long agonist or antagonist protocols. For long protocol, gonadotropin-releasing hormone analogue (GnRHa) will be given for pituitary desensitization, on Day 2-3 of the menstrual cycle, they will undergo transvaginal ultrasound examination and serum E2 measurement. Human menopausal gonadotrophin (hMG) or recombinant FSH will started at 150-300 IU per day based on the antral follicle count, age of women and previous ovarian response, according to the standard operation procedures of the centre. Ovarian response was monitored by serial transvaginal scanning with or without hormonal monitoring. Further dosage adjustments will base on the ovarian response at the discretion of the clinicians in charge. For antagonist protocols, antagonist (cetritide0.25mg daily) will be given on the 6th day of ovarian stimulation until day of hcg priming.

When three leading follicles were ≥18 mm, hCG 10 000 IU or ovidrel 250 mg will be given to trigger final maturation of oocytes. Oocyte retrievals will be arranged around 36 h later.

4.2 Insemination Procedures

All semen samples were prepared by the conventional swim-up procedure. At2hr after oocyte retrieval, each matured oocyte will be inseminated with approximately 50,000-100,000 motile spermatozoa.

4.3. Assignment and masking

On the day of OPU, patients will be randomized after occyte pick up by a laboratory technician according to a computer generated randomization list in sealed envelopes into the shorter incubation group or the control group. Until the completion of the whole study, both the patients and the clinicians were blinded to the group assigned.

Control arm Women who allocated to the control arm, all the oocytes will be exposed to spermatozoa for 20 hours, and checked for fertilization on day 1 (20 hours) after denuding

Intervention arm For those allocated to the intervention arm, all the oocytes will be exposed to spermatozoa for 2 hours and gently wash through two organ dishes containing 1.5 ml of equilibrated medium, and then transferred to the corresponding microdroplet of equilibrated fresh medium. Surrounding cumulus cell will be retained, not removed from the ooctyes.

4.4 Fertilization and Embryo Evaluation Both groups of oocytes will be decoronated and checked for the presence of two pronuclei and two polar bodies to confirm fertilization. All other outcomes (i.e., no fertilization, one pronucleus, polyspermia, degeneration) were also recorded.

Embryo morphology will be assessed every day of culture. Embryos will be scored according to the following criteria. Briefly, embryos are classified as: gradeA, no cellular fragmentation; grade B, <20% fragmentation; grade C, 20% to 50% fragmentation; and grade D, >50% fragmentation. The number of blastomeres per embryo was also recorded. Grade A and B embryos constituted the "good quality embryo".

The transfer is performed by the team clinician with a maximum of 2 embryos being replaced according to the standard protocol under transabdominal ultrasound guidance. Luteal phase support is given at the discretion of the physician.

4.5 Follow up strategy:

A pregnancy test will be carried out 2 weeks after embryo transfer in both arms. All women who have a positive pregnancy test 2 weeks after a fresh embryo transfer will undergo a transvaginal ultrasound scan after a further 5 weeks to identify the presence of a gestation sac with a fetal heart signifying an ongoing pregnancy.

Data on all pregnancy outcomes including early pregnancy losses such as miscarriage or ectopic pregnancy will be collected.

In order to achieve consistency with respect to the collection of outcome, standardised case report forms (CRF) will be completed for each woman at each centre. These CRFs will include details on treatment received, pregnancy outcomes, complications in pregnancy, mode of delivery and birth outcomes.

Statistics

5.1 Analysis plan: Demographic factors and clinical characteristics collected as part of baseline data collection will be summarised with counts (percentages) for categorical variables, mean (standard deviation [SD]) for normally distributed continuous variables, or median (interquartile [IQR] or entire range) for other continuous variables.

Outcomes for participants will be analysed in the groups to which they are assigned regardless of deviation from the protocol or treatment received (intention-to-treat). Comparative statistical analysis will entail calculating the relative risk (RR) (95% CI) for the primary outcome (99% CIs for all dichotomous secondary outcomes), the mean difference (99% CI) for normally distributed continuous secondary outcomes, or the median difference (99% CI) for skewed continuous variables.

All analyses will adjust for the minimisation factors to account for the correlation between treatment groups introduced by balancing the randomisation (which forces outcomes between treatment arms to be similar apart from any treatment effect).

Adjusted risk ratios will be estimated using a log binomial regression model, or using a log Poisson regression model with a robust variance estimator if the binomial model fails to converge. Linear regression will be used for normally distributed outcomes and quantile regression for skewed continuous variables.

Pre-specified subgroup analyses will include Cleavage versus blastocyst stage transfer.

6. Sample size estimation:

The average live birth rate in our center from 2010-2012 was 30% per transfer. According to recent published Meta analysis[11],brief co-incubation of gametes was associated with significantly higher rates of ongoing pregnancy (RR: 1.73, 95%CI: 1.27-2.33) than standard insemination.

Assuming live birth in the treatment group =50% (increase by 70%); with 90% power and a two-sided 5% level of statistical significance, we will need to recruit 124 women in each arm. To account for 10% loss to follow up, we will recruit 140 subjects in each group or 280 subjects for the whole study.

7. Assessment of safety

Recults from recent published Meta analysis[11,12] showed the rates of normal fertilization, good quality embryos and polyspermy were not significantly different with short time incubation of gametes compared with standard insemination. Thus, there should be no major safety concern in this study.

8. Direct access to source data / documents:

Trial-related monitoring, audits, IRB review and regulatory inspections are allowed.

9. Quality control and quality assurance

Patients will be managed by the listed investigators who have adequate experience in managing assisted reproduction treatments. A Trial steering committee will be formed which will oversee the conduct of the trial.

10. Ethics

Written consent will be obtained from all patients. The patient information sheet and consent forms in English and Chinese are enclosed. Ethics approval will be obtained from the Institutional Review Board, Shanghai first Maternity and Infant health hospital Hospital.

11. Data Handling and record keeping

All data will be stored for three years. A designated research nurse will be responsible for data management including data coding, monitoring and verification.

12. Financing and insurance

The study will be funded by MerckSerono China Research Fund for Fertility Experts.

13. Publication policy

The findings of this study will be submitted for consideration for publication in peer-reviewed scientific journal.

14. Supplements

The study will be conducted in compliance with the Declaration of Helsinki and Good Clinical Practice (ICH-GCP)

ELIGIBILITY:
Inclusion Criteria:

* Women under 42 years of age
* Any indications for conventional insemination such as tubal, endometriosis, unexplained and mild male factor
* Written informed consent

Exclusion Criteria:

* Women using donor eggs/donor sperm
* Women with abnormal uterine cavity shown on hysterosalpingogram or saline infusion sonogram
* Women with hydrosalpinges shown on scanning and not corrected treated
* Husband with severe oligospermia or azospermia or teraspermia (nomal morphology<5%)
* Previous fertilization failure for conventional insemination in the past (fertilization rate<30%)

Max Age: 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
live birth rate. | 1 year
  Number of live birth per transfer cycle

SECONDARY OUTCOMES:
Miscarriage rate | 1 year
Clinical pregnancy rates | 1 year
Normal fertilization rate | 1 year
polyspermy rate(>=3PN) | 1 year
Cleavage rate | 1 year
Implantation rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai first Maternity and Infant health hospital, Tong Ji University, Shanghai, China

REFERENCES:
- [Background] Waldenstrom U, Hamberger L, Nilsson L, Ryding M. Short-time sperm-egg exposure to prevent zona hardening. J Assist Reprod Genet 1993;10:190
- [Background] Wassarman PM. Fertilization in mammals. Sci Am. 1988 Dec;259(6):78-84. doi: 10.1038/scientificamerican1288-78. No abstract available. PMID 2849808
- [Background] Gianaroli L, Fiorentino A, Magli MC, Ferraretti AP, Montanaro N. Prolonged sperm-oocyte exposure and high sperm concentration affect human embryo viability and pregnancy rate. Hum Reprod. 1996 Nov;11(11):2507-11. doi: 10.1093/oxfordjournals.humrep.a019149. PMID 8981145
- [Background] Kattera S, Chen C. Short coincubation of gametes in in vitro fertilization improves implantation and pregnancy rates: a prospective, randomized, controlled study. Fertil Steril. 2003 Oct;80(4):1017-21. doi: 10.1016/s0015-0282(03)01154-3. PMID 14556826
- [Background] Lundqvist M, Johansson U, Lundkvist O, Milton K, Westin C, Simberg N. Reducing the time of co-incubation of gametes in human in-vitro fertilization has no beneficial effects. Reprod Biomed Online. 2001;3(1):21-24. doi: 10.1016/s1472-6483(10)61959-1. PMID 12513887
- [Background] Chen C, Kattera S. Rescue ICSI of oocytes that failed to extrude the second polar body 6 h post-insemination in conventional IVF. Hum Reprod. 2003 Oct;18(10):2118-21. doi: 10.1093/humrep/deg325. PMID 14507831
- [Background] Zhang XD, Liu JX, Liu WW, Gao Y, Han W, Xiong S, Wu LH, Huang GN. Time of insemination culture and outcomes of in vitro fertilization: a systematic review and meta-analysis. Hum Reprod Update. 2013 Nov-Dec;19(6):685-95. doi: 10.1093/humupd/dmt036. Epub 2013 Aug 2. PMID 23912477
- [Background] Huang Z, Li J, Wang L, Yan J, Shi Y, Li S. Brief co-incubation of sperm and oocytes for in vitro fertilization techniques. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD009391. doi: 10.1002/14651858.CD009391.pub2. PMID 23633370
- [Result] Gianaroli L, Cristina Magli M, Ferraretti AP, Fiorentino A, Tosti E, Panzella S, Dale B. Reducing the time of sperm-oocyte interaction in human in-vitro fertilization improves the implantation rate. Hum Reprod. 1996 Jan;11(1):166-71. doi: 10.1093/oxfordjournals.humrep.a019011. PMID 8671180
- [Result] Dirnfeld M, Bider D, Koifman M, Calderon I, Abramovici H. Shortened exposure of oocytes to spermatozoa improves in-vitro fertilization outcome: a prospective, randomized, controlled study. Hum Reprod. 1999 Oct;14(10):2562-4. doi: 10.1093/humrep/14.10.2562. PMID 10527987
- [Result] Dirnfeld M, Shiloh H, Bider D, Harari E, Koifman M, Lahav-Baratz S, Abramovici H. A prospective randomized controlled study of the effect of short coincubation of gametes during insemination on zona pellucida thickness. Gynecol Endocrinol. 2003 Oct;17(5):397-403. doi: 10.1080/09513590312331290288. PMID 14710587
- [Result] Barraud-Lange V, Sifer C, Pocate K, Ziyyat A, Martin-Pont B, Porcher R, Hugues JN, Wolf JP. Short gamete co-incubation during in vitro fertilization decreases the fertilization rate and does not improve embryo quality: a prospective auto controlled study. J Assist Reprod Genet. 2008 Jul;25(7):305-10. doi: 10.1007/s10815-008-9240-3. Epub 2008 Aug 1. PMID 18670871
- [Derived] Chen ZQ, Wang Y, Ng EHY, Zhao M, Pan JP, Wu HX, Teng XM. A randomized triple blind controlled trial comparing the live birth rate of IVF following brief incubation versus standard incubation of gametes. Hum Reprod. 2019 Jan 1;34(1):100-108. doi: 10.1093/humrep/dey333. PMID 30445454